CLINICAL TRIAL: NCT03803553
Title: Early Identification and Treatment of Occult Metastatic Disease in Stage III Colon Cancer
Brief Title: Identification and Treatment Of Micrometastatic Disease in Stage III Colon Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Stand Up To Cancer (Other)
Responsible Party: Principal Investigator, Aparna Parikh, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-397
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colon Cancer; Stage III Colon Cancer
Keywords: Metastatic colon Cancer; Stage III Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — IFL protocol; Watchful Waiting; Nivolumab; encorafenib; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- ctDNA-POSITIVE: FOLFIRI Protocol (Experimental): Pre-screening evaluation, including tumor assessment, tumor sequencing and blood tests. If these tests show that the participant is eligible to participate in the research study . The participant will be randomized into 1 of 3 groups : ctDNA-Positive: Folfiri or ctDNA-Positive: Active Surveillance or ctDNA Negative: Active Surveillance
  - ctDNA-POSITIVE: FOLFIRI Protocol
  * FOLFIRI chemotherapy via intravenous infusion on days 1-3 of each cycle. Cycle is 14 days long. This will occur for up to 12 cycles (24 weeks).
  * infusions will consist of the drugs
  * 5-Fluorouracil
  * Irinotecan
  * Leucovorin
  Interventions: Drug: FOLFIRI Protocol
- ctDNA-POSITIVE: ACTIVE SURVEILLANCE (Active Comparator): Pre-screening evaluation, including tumor assessment, tumor sequencing and blood tests. If these tests show that the participant is eligible to participate in the research study . The participant will be randomized into 1 of 3 groups : ctDNA-Positive: Folfiri or ctDNA-Positive: Active Surveillance or ctDNA Negative: Active Surveillance
  -- Active surveillance.
  * Observation and monitoring with imaging (every 3 months), tumor markers, and ctDNA draws every 1 month for the initial 6 months.
  * After 6 months, followed with ctDNA, tumor markers, and scans every 3 months for the first 3 years and every 6 months thereafter.
  Additional scans and tumor markers will be at the discretion of the clinician. .
  Interventions: Other: ACTIVE SURVEILLANCE
- ctDNA-NEGATIVE: ACTIVE SURVEILLANCE (Active Comparator): Pre-screening evaluation, including tumor assessment, tumor sequencing and blood tests. If these tests show that the participant is eligible to participate in the research study . The participant will be randomized into 1 of 3 groups : ctDNA-Positive: Folfiri or ctDNA-Positive: Active Surveillance or ctDNA Negative: Active Surveillance
  - Observation and monitoring with imaging, tumor markers, and ctDNA collections every 3 months for the first 3 years and every 6 months thereafter.
  Additional scans and tumor markers will be at the discretion of the clinician
  Interventions: Other: ACTIVE SURVEILLANCE
- ctDNA-POSITIVE MSI-H: NIVOLUMAB (Experimental): Pre-screening evaluation, including tumor assessment, tumor sequencing and blood tests.
  If these tests show that the participant is eligible to participate in the research study and is ctDNA positive and MSI-H, the participant will not be randomized and will be placed into the group: ctDNA positive, MSI-H: Nivolumab
  -ctDNA-Positive, MSI-H: Nivolumab Protocol
  * Nivolumab treatment via intravenous infusion on day 1 of each cycle. Cycle is 28 days long. This will occur for up to 12 cycles (48 weeks).
  * infusions will consist of the drug Nivolumab
  Interventions: Drug: Nivolumab Protocol
- ctDNA-POSITIVE BRAF Mutant: ENCORAFENIB/BINIMETINIB/CETUXIMAB (Experimental): Pre-screening evaluation, including tumor assessment, tumor sequencing and blood tests.
  If these tests show that the participant is eligible to participate in the research study and is ctDNA positive and has a BRAF mutation, the participant will not be randomized and will be placed into the group: ctDNA positive, BRAF mutant: Encorafenib/Binimetinib/Cetuximab
  -ctDNA-Positive, MSI-H: Encorafenib/Binimetinib/Cetuximab Protocol
  * Encorafenib/Binimetinib treatment is received orally every day and Cetuximab via intravenous infusion on day 1 of each cycle. Cycle is 14 days long. This will occur for up to 12 cycles (24 weeks).
  * infusions will consist of the drug Cetuximab
  Interventions: Drug: Encorafenib/Binimetinib/Cetuximab Protocol
- 6 Months Additional Trastuzumab and Pertuzumab (Experimental): Pre-screening evaluation, including tumor assessment, tumor sequencing and blood tests. Participants that are eligible to receive Trastuzumab and Pertuzumab will be placed in this HER2 cohort: ctDNA-positive & HER2 amplification and MSS Trastuzumab and Pertuzumab. Trastuzumab is received via intravenous administration, and Pertuzumab treatment is received intravenously by infusion. Cycle is 21 days. This will occur for up to 8 cycles.
  Interventions: Drug: Trastuzumab + Pertuzumab

INTERVENTIONS:
Drug: FOLFIRI Protocol — FOLFIRI cycle will be two weeks (14 days) long, with FOLFIRI administered on Days 1-3. Participants will receive up to 12 two-week cycles (for a total of 24 weeks) of FOLFIRI chemotherapy.
  Other Names: FOLinic acid-Fluorouracil-IRInotecan regimen
  Arms: ctDNA-POSITIVE: FOLFIRI Protocol
Other: ACTIVE SURVEILLANCE — Will be followed with observation and monitoring with imaging, tumor markers, and ctDNA collections
  Arms: ctDNA-NEGATIVE: ACTIVE SURVEILLANCE; ctDNA-POSITIVE: ACTIVE SURVEILLANCE
Drug: Nivolumab Protocol — Nivolumab cycle will be four weeks (28 days) long, with Nivolumab administered on day 1. Participants will receive up to 12 four-week cycles (for a total of 48 weeks) of Nivolumab treatment.
  Other Names: Nivolumab
  Arms: ctDNA-POSITIVE MSI-H: NIVOLUMAB
Drug: Encorafenib/Binimetinib/Cetuximab Protocol — Encorafenib/Binimetinib will be taken orally every day and Cetuximab will be administered intravenously on day 1 of each cycle. Cycles are 14 days long. Participants will receive up to 12 two-week cycles (for a total of 24 weeks) of Encorafenib/Binimetinib/Cetuximab.
  Other Names: Enco/Bini/Cetux
  Arms: ctDNA-POSITIVE BRAF Mutant: ENCORAFENIB/BINIMETINIB/CETUXIMAB
Drug: Trastuzumab + Pertuzumab — Trastuzumab (Herceptin) is received by intravenous administration and Pertuzumab is received intravenously by infusion on Day 1 of each cycle. Cycles are 21 days long. Participants will receive up to 8 cycles of Trastuzumab and Pertuzumab.
  Other Names: Herceptin
  Arms: 6 Months Additional Trastuzumab and Pertuzumab

SUMMARY:
This research study is comparing two standard of care treatment options based on blood test results for participants who have metastatic colon cancer.

The names of the potential treatments involved in this study are:

* Active surveillance
* FOLFIRI treatment
* Nivolumab treatment
* Encorafenib/Binimetinib/Cetuximab treatment
* Trastuzumab + Pertuzumab

DETAILED DESCRIPTION:
The FDA (the U.S. Food and Drug Administration) has approved FOLFIRI, comprised of Irinotecan, Leucovorin, and 5-Fluorouracil, as a treatment option for metastatic colon cancer in the Stage IV setting.

* After diagnosis and surgical removal of tumors, individuals with metastatic colon cancer commonly receive what is called adjuvant chemotherapy treatment, commonly utilizing treatment plans called FOLFOX, CAPOX, or therapy with 5-Fluorouracil.
* If all the cancer is not killed, the investigators may be able to detect tumor in the blood called circulating tumor DNA (ctDNA). This is genetic material unique to metastatic colon cancer that may be present in the blood stream, and it can be identified through a ctDNA blood test. If ctDNA is present in the blood stream, it is commonly called micro-metastatic disease (meaning disease that can't be seen detected by CT scans but may be there in the blood). Cancer researchers believe that ctDNA in the blood stream may be an indicator that cancer is more likely to recur.
* After initial adjuvant chemotherapy, it is standard for individuals to begin active surveillance, where they do not receive further treatment but instead undergo frequent tumor imaging scans to see if their cancer is stable, growing, or coming back. The investigators plan to see if additional therapy, where FOLFIRI (comprised of Irinotecan, Leucovorin, and 5-Fluorouracil) is administered can decrease recurrence. Typically, FOLFIRI is given when the disease is visibly recurrent.

  * In addition, the investigators plan to include study groups of adjuvant nivolumab treatment and adjuvant Encorafenib/Binimetinib/Cetuximab treatment to see if these treatments can decrease recurrence. The FDA has not approved either of these as a treatment options for metastatic colon cancer in the Stage IV setting.
  * Patients who have a greater than normal number of genetic markers called microsatellites are called MSI-H. Because tumor cells with these features tend to have more genetic mutations than tumor cells without them, they are more likely to be recognized by the immune system. Nivolumab is an anti-PD-1 antibody. It works by attaching to and blocking a molecule called PD-1. PD-1 is a protein that is present on different types of cells in your immune system and controls parts of your immune system by shutting it down. Antibodies that block PD-1 can potentially prevent PD-1 from shutting down the immune system, thus potentially allowing immune cells to recognize and destroy cancer cells.
  * Encorafenib in combination with binimetinib and cetuximab is one of the first effective regimens to target the BRAF V600E-mutation in colon cancer. When this mutation is present, it switches on pathway called the MAPK pathway which stimulates cell division and leads to uncontrolled cell growth. Encorafenib, binimetinib and cetuximab target different parts of this important signaling pathway in tumor cells with this mutation and slows down their growth and communication

However, in this research study, the investigators are

* determining whether there are differences in cancer recurrence in ctDNA positive participants treated with additional therapy versus put on active surveillance.
* determining whether there are differences in health in ctDNA positive participants treated with additional therapy versus put on active surveillance.
* examining whether patients who undergo further therapy experience changes in the ctDNA levels.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed resected Stage III adenocarcinoma of the colon. Any T [Tx, T1, T2, T3, or T4-], N1-2M0.
* Participants must have completely resected disease. In patients with tumor adherent to adjacent structures, en block RO resection must be documented.
* Entire tumor must be in the colon (rectal involvement is excluded).
* Participants must have completed standard adjuvant chemotherapy per the discretion of the treating physician. Standard therapy includes FOLFOX, CAPOX, or therapy with 5FU analog alone will be permitted if it constitutes appropriate standard therapy in the opinion of the treating physician.
* Participants must not have received prior neoadjuvant chemotherapy.
* Age ≥18 years.
* ECOG performance status ≤1.
* Life expectancy of greater than 3 months.
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/ mcL
  * total bilirubin within normal institutional limits. For patients with Gilbert's syndrome, total bilirubin must be ≤ 2 and documented as elevated indirect bilirubin.
  * AST(SGOT)/ALT(SGPT) ≤3 (AST) or ≤ 3 (ALT) × institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥40 mL/min/1.73 m2 for participants with creatinine levels above institutional normal by Cockroft-Gault formula.
* In order to be eligible for the ctDNA positive cohort, women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG).
* The effects on the developing human fetus are unknown. For this reason and because 5FU, Capecitabine, Oxaliplatin, Irinotecan, Leucovorin, Nivolumab, and Cetuximab are known to be teratogenic, in order to be eligible for the ctDNA positive cohort, females of child-bearing potential (FOCBP) and males must be willing to abstain from heterosexual activity or use 2 forms of effective contraception (fail rate of less than 1% per year, hormonal or barrier method of birth control) from time of informed consent until 5 months (FOCBP) and 7 months (males) after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women who are not of childbearing potential, ie, who are postmenopausal or surgically sterile as well as azoospermic men, do not require contraception.
* Participants must have documentation of microsatellite instability status. Testing by NGS, PCR based assessment and Immunohistochemistry (IHC) are acceptable. Presence of deficient (d) DNA mismatch repair (dMMR) may be assessed by IHC for MMR protein expression (MLH1, MSH2, MSH6, PMS2) where loss of one or more proteins indicated dMMR. This may be done locally.
* Participant's circulating tumor DNA (ctDNA) assay (Guardant Reveal-Guardant Health) must satisfy assay specific quality control metrics to generate a result.
* In order to be eligible for the ctDNA positive cohort, patient must be ctDNA positive following adjuvant therapy using the CLIA certified Guardant Reveal assay. ctDNA positive will be defined as positive based on having a tumor derived signal in the cfDNA that passes calling threshold ("ctDNA detected").
* Ability to understand and the willingness to sign a written informed consent document.

Trastuzumab and Pertuzumab Specific Inclusion Criteria for HER2 cohort

* HER2 overexpression/amplification as shown by NGS sequencing, IHC/FISH or Tumor with 3+ by IHC or 2+ by IHC and HER2/cep17 ratio >2 by FISH.
* AST(SGOT) ≤ 1.25 and ALT(SGPT) ≤ 1.25 × institutional upper limit of normal
* Participants of childbearing potential must use effective contraceptive methods during and for 7 months after the last dose of HER2-targeted therapy
* History of other malignancies within the 5 years prior to study registration, except for the following: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinomas of the skin (*malignancies occurring more than 5 years prior to study entry are permitted if curatively treated with surgery alone).
* LVEF ≥ 55% measured by echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA) within 12 weeks of treatment start.

Exclusion Criteria:

* Patients who are receiving additional investigational therapy or on another investigational protocol
* Patients who have confirmed metastatic disease per CT.
* Patients who are unable to get any standard adjuvant therapy
* Patients who have received more than 6 months of standard adjuvant therapy at the time of study entry.
* With the exception of standard of care adjuvant therapy, patient received anticancer therapy including chemotherapy, immunotherapy, or antineoplastic biologic therapy (e.g., cetuximab, bevacizumab etc.), within 30 days prior to start of study treatment.
* Patients who are MSI-high or have a BRAF V600E mutation are excluded from Arm 1 (FOLFIRI) and Arm 2 (Active Surveillance).
* Patients with a BRAFV600E mutation and who are MSI-high are excluded from Arm 5 (ENCO/BINI/CETUX).
* Has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* (ctDNA positive cohort only). Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 6 months for woman and 6 months for men, after the last dose of trial treatment.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin and squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has an active infection requiring systemic therapy.

Nivolumab Specific Inclusion Criteria for MSI-H Cohort:

* Must have documentation of microsatellite instability status. NGS, PCR based assessment and Immunohistochemistry (IHC) are acceptable. Presence of deficient (d) DNA mismatch repair (dMMR) may be assessed by IHC for MMR protein expression (MLH1, MSH2, MSH6, PMS2) where loss of one or more proteins indicated dMMR. This may be done locally.
* Patients must have detectable ctDNA (Guardant Reveal assay) post standard adjuvant therapy in order to be in this cohort.

Nivolumab Specific Exclusion Criteria for MSI-H Cohort:

* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other forms of immunosuppressive therapy within 7 days prior to the first dose of nivolumab treatment. Subject requiring systemic steroids are excluded from the trial. The use of physiologic doses of corticosteroids may be approved after discussion with the sponsor.
* Has a known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to nivolumab or any of is excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Patients that require supplemental oxygen are excluded.
* Patients who are known HIV+ positive are eligible if their CD4+ count is ≥ 350/μL for at least 3 months and they have an undetectable viral load. In addition, patient must be currently receiving Highly Active Antiretroviral Therapy (HAART) and have been on therapy for at least 3 months prior to study entry, under the care of an Infectious Diseases specialist. Patients should have no history of an AIDS-defining opportunistic infection.
* Patients known hepatitis B and hepatitis C must be under the care of viral hepatitis expert consultant. Patients with hepatitis B are required to be treated with anti-HBV treatment (e.g., entecavir) and have an HBV viral load <100 IU/mL. Patients with hepatitis C need to have received prior and/or ongoing hepatitis C treatment.
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Encorafenib, binimetinib, and cetuximab Specific Inclusion Criteria for BRAF mutant Cohort

* Presence of BRAFV600E in tumor tissue previously determined by IMPACT at any time prior to Screening.
* Patients must have detectable ctDNA (Guardant Health LUNAR assay) post standard adjuvant therapy in order to be in this cohort.
* Participants must have normal organ, marrow, and hematologic function as defined below:

  * Hemoglobin ≥9 g/dL (5.58 mmol/L)
  * Total bilirubin ≤ 1.5 (25.65 μmol/L)
  * Platelets ≥100,000/μL

Encorafenib, binimetinib, and cetuximab Specific Exclusion Criteria for BRAF V600E mutant Cohort:

* Patients with a BRAFV600E mutation and who are MSI-H are excluded from Arm 5 (ENCO/BINI/CETUX)
* Prior therapy with a BRAF inhibitor (e.g., encorafenib, dabrafenib, vemurafenib) and/or a MEK inhibitor (e.g., binimetinib, trametinib, cobimetinib).
* Known hypersensitivity or contraindication to any component of binimetinib or encorafenib or their excipients.
* The patient has a history of allergic reactions attributed to compounds of chemical or biologic composition similar to those of cetuximab, or has red meat allergy or tick bit history.
* Inability to swallow and retain study drug.
* Participants who have undergone major surgery (e.g., in-patient procedures) ≤ 6 weeks prior to start of study treatment or who have not recovered from side effects of such procedure.
* Participants who have had radiotherapy ≤ 14 days prior to start of study treatment or who have not recovered from side effects of such procedure. Note: Palliative radiation therapy must be complete 7 days prior to the first dose of study treatment.
* Patient has not recovered to ≤ Grade 1 from toxic effects of prior therapy before starting study treatment.

Note: Stable chronic conditions (≤ Grade 2) that are not expected to resolve (such as neuropathy, myalgia, alopecia, prior therapy-related endocrinopathies) are exceptions and may enroll.

* Impaired cardiovascular function or clinically significant cardiovascular disease including, but not limited to, any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stenting) < 6 months prior to Screening;
  * Congestive heart failure requiring treatment (New York Heart Association Grade ≥ 2);
  * Left ventricular ejection fraction (LVEF) < 50% as determined by MUGA or ECHO;
  * Uncontrolled hypertension defined as persistent systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg despite current therapy;
  * History or presence of clinically significant cardiac arrhythmias (including resting bradycardia, uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia);
  * Triplicate average baseline QTc interval ≥ 480 ms.
* Impairment of gastrointestinal function or disease which may significantly alter the absorption of study drug (e.g., active ulcerative disease, uncontrolled vomiting or diarrhea, malabsorption syndrome, small bowel resection with decreased intestinal absorption), or recent (≤ 3 months) history of a partial or complete bowel obstruction, or other conditions that will interfere significantly with the absorption of oral drugs.
* Known history of acute or chronic pancreatitis.
* Concurrent neuromuscular disorder that is associated with elevated CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
* History or current evidence of RVO or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes); history of retinal degenerative disease.
* Current use of a prohibited medication (including herbal medications, supplements, or foods), as described in Section 5.5, or use of a prohibited medication ≤ 1 week prior to the start of study treatment.
* History of thromboembolic or cerebrovascular events ≤ 12 weeks prior to the first dose of study treatment. Examples include transient ischemic attacks, cerebrovascular accidents, hemodynamically significant (i.e. massive or sub-massive) deep vein thrombosis or pulmonary emboli.

Note: Patients with either deep vein thrombosis or pulmonary emboli that does not result in hemodynamic instability are allowed to enroll as long as they are on a stable dose of anticoagulants for at least 4 weeks.

Note: Patients with thromboembolic events related to indwelling catheters or other procedures may be enrolled.

* Concurrent or previous other malignancy within 2 years of study entry, except adequately treated basal or squamous cell skin cancer, prostate intraepithelial neoplasm, carcinoma in-situ of the cervix, Bowen's disease and Gleason 6 prostate cancer.
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Evidence of Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) infection. Note: Patients with laboratory evidence of cleared HBV or HCV infection may be enrolled.

Note: Patients with no prior history of HBV infection who have been vaccinated against HBV and who have a positive antibody against hepatitis B surface antigen as the only evidence of prior exposure may be enrolled.

Trastuzumab and Pertuzumab Specific Exclusion Criteria for HER2 cohort

* Serious cardiac illness or medical conditions including but not confined to:

  * History of NCI CTCAE v5.0 Grade ≥ 3 symptomatic congestive heart failure (CHF) or New York Heart Association (NYHA) Class ≥ II
  * High-risk uncontrolled arrhythmias ie, atrial tachycardia with a heart rate ≥ 100/min at rest, significant ventricular arrhythmia (ventricular tachycardia) or higher-grade AV-block (second degree AV-block Type 2 [Mobitz 2] or third degree AV-block)
  * Serious cardiac arrhythmia or severe conduction abnormality not controlled by adequate medication
  * Angina pectoris requiring anti-anginal medication.
  * Evidence of myocardial infarction within 12 months prior to enrollment
  * Clinically significant valvular heart disease
  * Evidence of transmural infarction on electrocardiogram (ECG)
  * Poorly controlled hypertension (eg, systolic > 180 mm Hg or diastolic > 100 mm Hg).
  * History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias, such as structural heart disease (e.g., severe left ventricular systolic dysfunction [LVSD], left ventricular hypertrophy), coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing), clinically significant electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia), or family history of sudden unexplained death or long QT syndrome
* High risk patients who have received chemoprevention drugs in the past are not allowed to enroll in the study.
* Concurrent anti-cancer treatment in another investigational trial, including hormone therapy, bisphosphonate therapy and immunotherapy.
* Other concurrent serious diseases that may interfere with planned treatment including severe pulmonary conditions/illness (e.g., infections or poorly controlled diabetes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 5 years
  Disease-free survival (DFS) between ctDNA-positive patients treated with additional treatment of FOLFIRI and ctDNA-positive patients who are untreated
Clearance rate of ctDNA | 7 Months
  Compare the clearance rate of ctDNA in ctDNA-positive patients between patients treated with additional treatment of FOLFIRI and those who are untreated

SECONDARY OUTCOMES:
Overall Survival (OS) Rate | 5 years
  Overall survival (OS) between ctDNA-positive patients treated with additional adjuvant therapy (Arm 1) and ctDNA-positive patients who are untreated (Arm 2)
Clearance rate of ctDNA of Arm 4: Nivolumab Treatment | 13 months
  Determine clearance rate of ctDNA-positive patients treated with nivolumab in an exploratory MSI/mismatch repair deficient cohort
Disease-free survival (DFS) of Arm 4: Nivolumab Treatment | 5 years
  Determine the disease-free survival (DFS) of ctDNA-positive patients treated with nivolumab in an exploratory MSI/mismatch repair deficient cohort
Clearance rate of ctDNA of Arm 5: Encorafenib/Binimetinib/Cetuximab Treatment | 7 months
  Determine the clearance rate of ctDNA-positive patients treated with encorafenib, binimetinib, and cetuximab in an exploratory BRAF V600E cohort.
Disease-free survival (DFS) of Arm 5: Encorafenib/Binimetinib/Cetuximab Treatment | 5 years
  Determine the disease-free survival DFS of ctDNA-positive patients treated with encorafenib, binimetinib, and cetuximab, in an exploratory BRAF V600E cohort.
ctDNA clearance as Marker | 13 Months
  Examine the correlation of ctDNA clearance as a surrogate marker for disease burden
Lead time to recurrence | 5 years
  Compare lead time to recurrence and sensitivity of predicting recurrence between ctDNA and tumor markers
Disease-free survival (DFS) of Arm 6: Herceptin/Perjeta | 5 years
  Determine the DFS ctDNA-positive patients treated Herceptin/Perjeta
Clearance rate of Arm 6: Herceptin/Perjeta | 7 months
  Determine the clearance rate of ctDNA-positive patients treated Herceptin/Perjeta

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Parikh, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation